CLINICAL TRIAL: NCT07239713
Title: Clinical Effects of Ringers Lactate Versus Sterofundin/Plasmalyte Solution in Surgical Adult Patients With Sepsis; a Comparative Study in ICU Patients
Brief Title: Clinical Effects of Ringers Lactate Versus Sterofundin/ Plasmalyte Solution in Patients With Sepsis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CMH Lahore Medical College and Institute of Dentistry (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 563/2024
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Post Abdominal Surgery; Sepsis Abdominal
Keywords: Fluid therapy; Abdominal Surgery; Postoperative; Sepsis
MeSH Terms: conditions — Intraabdominal Infections; Sepsis | interventions — sterofundin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ringer's Lactate Group (Active Comparator): This group will receive RInger's Lactate as maintenance fluid.
  Interventions: Other: Ringer's Lactate Crystalloid Solutions
- Steroundin Group (Experimental): This group will receive Sterofundin as maintenance fluid.
  Interventions: Other: Sterofundin (Bolus of crystalloids)

INTERVENTIONS:
Other: Ringer's Lactate Crystalloid Solutions — A balanced crystalloid solution containing sodium, potassium, calcium, chloride, and lactate as a buffer.
  Used at a standard maintenance rate for adult postoperative patients.
  Arms: Ringer's Lactate Group
Other: Sterofundin (Bolus of crystalloids) — A balanced, multi-electrolyte crystalloid solution containing acetate and malate as buffers instead of lactate.
  Designed to more closely match plasma electrolyte composition, with a lower chloride concentration than RL.
  Arms: Steroundin Group

SUMMARY:
The goal of this clinical trial is to compare the clinical effects of using Ringer's Lactate and Sterofundin/ Plasmalyte as maintenance fluids in adult patients who have undergone abdominal surgery and are septic.

The primary outcome will be the change in serum lactate levels. Secondary outcomes will include renal function parameters, qSOFA scores, and the incidence of postoperative complications within the first 72 hours following surgery.

DETAILED DESCRIPTION:
The goal of this clinical trial is to compare the clinical effects of using Ringer's Lactate and Sterofundin/PlasmaLyte as maintenance fluids in adult patients who have undergone abdominal surgery and are septic.

The primary outcome will be the change in serum lactate levels. Secondary outcomes will include renal function parameters, qSOFA scores, and the incidence of postoperative complications within the first 72 hours following surgery.

The main questions it aims to answer are:

1. Does the choice of fluid produce different outcomes in this patient population?
2. If yes, then which fluid produces better outcomes?

Enrolled patients will be randomly assigned Ringer's Lactate or Sterofundin for intravenous infusion. The volume, infusion rate and additive content will be determined by the treating clinicians. The intervention will last for 72 hours after patients' enrolment.

ELIGIBILITY:
Inclusion Criteria:

* Underwent Abdominal Surgery and postoperative length of stay is more than 24 hours
* ASA 1 to 4
* Diagnosis of sepsis (qSOFA score 2 or more)

Exclusion Criteria:

* Patients with Renal failure/hepatic failure/severe metabolic acidosis
* Patients requiring renal replacement therapy prior to enrolment
* Patients with suspected poisoning
* Pregnant women
* Patients having solitary kidney

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
serum lactate | Samples will be collected at baseline (preoperatively or immediately postoperatively) and at predefined intervals during the postoperative period (e.g., 24 and 48 hours after surgery).
  Measurement: Serum lactate levels will be measured from blood samples.
  Method: Standard laboratory assays will be used to quantify lactate concentration.
  Purpose: To assess the effect of maintenance fluids (Ringer's Lactate vs. Sterofundin) on lactate clearance and tissue perfusion in septic adult patients following abdominal surgery.
  Units: mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Syed A Jafri, MBBS, Study Chair — Combined military hospital lahore
Locations (1):
- Combined Military Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No